CLINICAL TRIAL: NCT06055777
Title: A Randomized, Double-blind, Placebo-controlled Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics of SZEY-2108 Administreated as Single and Repeated Intravenous Doses in Chinese Healthy Subjects
Brief Title: Study of the Safety, Tolerability, and PK of SZEY-2108 Administered Intravenously to HVs in SAD and MAD Cohorts
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to the termination criteria for dose escalation in the clinical protocol having been reached, this trial is terminated.
Sponsor: Suzhou Erye Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZEY-2108-I-01
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Infections
Keywords: Healthy volunteers; SZEY-2108
MeSH Terms: conditions — Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single intravenous doses of SZEY-2108 (Active Comparator): Single escalating doses of SZEY-2108
  Interventions: Drug: SZEY-2108 for injetion
- Single intravenous doses of placebo (Placebo Comparator): Single intravenous doses of placebo to match SZEY-2108
  Interventions: Drug: Placebo
- Multiple intravenous doses of SZEY-2108 (Active Comparator): Multiple intravenous doses of SZEY-2108 at Q8h or Q6h on D1~D7 and on the morning of D8.
  Interventions: Drug: SZEY-2108 for injetion
- Multiple intravenous doses of placebo (Placebo Comparator): Multiple intravenous doses of placebo at Q8h or Q6h on D1~D7 and on the morning of D8.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SZEY-2108 for injetion — Part1（Single-dose intravenous infusion dose-escalation trial）:100mg，200mg，500mg, 1000mg, 2000mg，4000mg and the dose of last cohort to be determined. Single intravenous doses on D1；Part 2（Multi-dose intravenous infusion dose-escalation trial）：1000mg at Q8h，2000mg at Q8h, and one dose level of 1000mg, 1500mg or 2000mg at Q6h. Multiple intravenous doses of SZEY-2108 at Q8h or Q6h on D1~D7 and on the morning of D8.
  Other Names: Novel monocyclic β-lactam antibiotics
  Arms: Multiple intravenous doses of SZEY-2108; Single intravenous doses of SZEY-2108
Drug: Placebo — Part1（Single-dose intravenous infusion dose-escalation trial）:250mL/500mL，Single intravenous doses on D1；Part 2（Multi-dose intravenous infusion dose-escalation trial）：250mL,Multiple intravenous doses of placebo at Q8h or Q6h on D1~D7 and on the morning of D8.
  Other Names: 0.9% Sodium Chloride Injection
  Arms: Multiple intravenous doses of placebo; Single intravenous doses of placebo

SUMMARY:
This phase 1 study was designed to evaluate the safety and tolerability of SZEY-2108 in single and multiple intravenous infusions, the pharmacokinetic profile of SZEY-2108 after single and multiple intravenous infusions, and the effect of exposure to SZEY-2108 after a single intravenous infusion on QT/QTc interval. Metabolites in each biological matrix (blood, urine, feces) and excretion characteristics (feces) after SZEY-2108 were analyzed.

DETAILED DESCRIPTION:
This is a first-in-human, randomized, double-blind, placebo-controlled study consisting of 2 parts. Part 1: Single-dose intravenous infusion dose-escalation trial. A total of 44 ~ 52 healthy adult subjects will be enrolled in Part 1 and they will be administrated with SZEY-2108 or placebo by single intravenous infusion. Part 1 consists of 7 cohorts: 100mg，200mg，500mg, 1000mg, 2000mg，4000mg and the dose of last cohort to be determined. Four subjects will be randomized to SZEY-2108 or placebo at a ratio of 1:1 in the 100mg cohort and eight subjects at a ratio of 3:1 in other each cohort. Time for intravenous infusion is 2h±5 min and it may be extended to 3 h±5 min if intolerance occur in 2000mg and 4000mg cohort.

Subjects will be randomised to receive an intravenous infusion of SZEY-2108 or placebo on the morning of D1, then they will still be hospitalised for safety, tolerability, pharmacokinetic and C-QTc assessment, and finally will discharge the Phase I clinical study centre after completion of all assessments at D3. They are required to return to the study centre at D7 for a safety follow-up visit.

Part 2: Multi-dose intravenous infusion dose-escalation trial According to results of Part 1, administration dose and dosing interval may be adjusted in Part 2.

Thirty healthy adult subjects will be enrolled in Part 2 and they will receive multiple doses of SZEY-2108 or placebo by intravenous infusion. Part 2 consists of 3 cohorts: 1000mg at Q8h，2000mg at Q8h, and one dose level of 1000mg, 1500mg or 2000mg at Q6h. Ten subjects will be randomized to SZEY-2108 or placebo at a ratio of 4:1 in each cohort. Time for intravenous infusion is 2h±5 min and it may be extended to 3 h±5 min if intolerance occur in 2000mg cohort.

Subjects will be randomized to receive an intravenous infusion of SZEY-2108 or placebo at Q8h or Q6h on D1~D7 and on the morning of D8. They will still be hospitalised for safety, tolerability and pharmacokinetic assessment, and finally will discharge the Phase I clinical study centre after completion of all assessments at D9 or D10 (for faecal retention group). Subjects are required to return to the study centre at D15 for a safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years at the time of screening;
* BMI between 19 and 28 kg/m2, and weight for males and females ≥ 50kg and 45kg, respectively;
* No clinical relevant abnormalities
* Sign informed consent

Exclusion Criteria:

* Any clinical significant illness
* Other medical or psychiatric may inappropriate for the study
* Past history of allergic conditions or current comorbid allergies
* Use of any prescription medications within 4 weeks prior to screening or use of any over-the-counter medications, herbs, supplements, and vitamins within 7 days prior to the use of the investigational drug;
* History of cigarette, alcohol or drug abuse
* Abnormal vital signs, such as blood pressure and pulse rate
* Abnormal examination results, such as 12-ECG, eGFR, ALT, AST and TBL
* Positive results of HBsAg, TPPA, HCV-Ab, or HIV-Ab
* Blood loss or donation > 400ml within 3 months prior to screening
* Pregant or breastfeeding females or subjects unwilling to contraception

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Safety of single and multiple ascending doses of SZEY-2108 | Part 1: From the time of signed consent through the end of study date which occurs on Day 7±1;Part 2: From the time of signed consent through the end of study date which occurs on Day 15±1
  Safety and tolerability as assessed through the determination and recording of the occurrence of AEs as well as by adverse changes in vital signs, ECG (e.g. QTc interval) parameters, and laboratory data.

SECONDARY OUTCOMES:
Assessment of Pharmacokinetic Parameter (plasma): Cmax measurement | In Part 1：0 to 24 hours post-dose on Day 1 ；In Part 2：0 to 24 hours post-dose on Days 1~7 and on the morning of D8 (varied intervals per cohort)
  Maximum plasma concentration (Cmax µg/mL) on Day 1 after single infusion , maximum plasma concentration at steady state (Css,max µg/mL) after multiple infusion.
Assessment of Pharmacokinetic Parameter (plasma): AUC | In Part 1：0 to 24 hours post-dose on Day 1 ；In Part 2：0 to 24 hours post-dose on Days 1~7 and on the morning of D8 (varied intervals per cohort)
  Area under the plasma concentration-time curve from zero extrapolated to infinity (AUC µg*h/mL) or AUC(0-last) in Part 1 on Day 1 after single infusion, area under the plasma concentration-time curve at steady state after multiple infusion (AUCss µg*h/mL).
Assessment of Pharmacokinetic Parameter (plasma): Tmax | In Part 1：0 to 24 hours post-dose on Day 1 ；In Part 2：0 to 24 hours post-dose on Days 1~7 and on the morning of D8 (varied intervals per cohort)
  The time to maximum observed concentration of study drug in plasma
Assessment of Pharmacokinetic Parameter (plasma): t1/2 | In Part 1：0 to 24 hours post-dose on Day 1 ；In Part 2：0 to 24 hours post-dose on Days 1~7 and on the morning of D8 (varied intervals per cohort)
  Terminal half-life (t1/2), on Day 1 after single infusion and at steady state after multiple infusion.
Assessment of Pharmacokinetic Parameter (plasma): CL | In Part 1：0 to 24 hours post-dose on Day 1 ；In Part 2：0 to 24 hours post-dose on Days 1~7 and on the morning of D8 (varied intervals per cohort)
  Systemic clearence (CL) on Day 1 after single infusion and at steady state after multiple infusion.
Assessment of Pharmacokinetic Parameter (urine): SZEY-2108 | In Part 1：Day1: baseline ,0 to 4, 4 to 8, 8 to 12 and 12 to 24h ；In Part 2：Day1: baseline,0 to 2, 2 to 4, 4 to 8, 8 to 12 and 12 to 24h.
  amount of SZEY-2108 excreted in urine
Quantitative relationship between blood concentration and QTc interval of SZEY-2108. | In Part 1：Before dosing (Baseline) through 24 hours after the dose on Day 1 （The dose groups of 100mg and 200mg were excluded）
  C-QTc will be analyzed using concentration-QT (cQT) modeling

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojie Wu, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No